CLINICAL TRIAL: NCT03546946
Title: Investigating Attention Patterns in Young People With Anxiety
Acronym: ATTN-ANX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 225926
Record Dates: First submitted 2017-10-20; First posted 2018-06-06 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Anxiety; Adolescent Behavior
Keywords: Attention; Anxiety; Adolescence
MeSH Terms: conditions — Anxiety Disorders; Adolescent Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gaze-Contingent Music Reward Training (Experimental): GCMRT for eight 20-minute sessions - twice per week over 4 weeks.
  Interventions: Behavioral: Gaze-Contingent Music Reward Training
- Control Training (Placebo Comparator): Passive viewing task with continuous music for eight 20-minute sessions - twice per week over 4 weeks.
  Interventions: Behavioral: Control Training
- No-Train Group (No Intervention): No active training.

INTERVENTIONS:
Behavioral: Gaze-Contingent Music Reward Training — Participants will hear their selected music track playing, dependent on their gaze location, when viewing a grid on neutral and negative faces.
  Arms: Gaze-Contingent Music Reward Training
Behavioral: Control Training — Participants will hear their selected music track playing, regardless of their gaze location, when viewing a grid on neutral and negative faces.
  Arms: Control Training

SUMMARY:
Adolescents with elevated anxiety have been found to direct their voluntary and involuntary attention more readily toward threatening stimuli, and spend more time dwelling upon that stimuli. Various computerised tasks have been developed to attempt to retrain these "attention biases" back away from threat.

This study will test a newly developed intervention, that uses (eye-tracking) methods to track the gaze of the individual. This intervention is called Gaze-Contingent Music Reward Training (GC-MRT), and is designed to re-train the individual away from dwelling upon threatening stimuli (emotional faces), using their favourite music to re-infornce this learning.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years of age upon study commencement
* Diagnosed generalised or social anxiety disorder (assessed by SCID)
* Informed written and witnessed consent

Exclusion Criteria:

* Psychosis
* Autism
* Learning difficulties
* Uncorrected abnormal vision
* Current use of SSRIs

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Estimated)
Dates: Start 2018-06-05 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety symtoms | Baseline and post-intervention (4 weeks), and at 3-month follow up.
  Change in anxiety symptoms from baseline at 4-weeks on the Kiddie Schedule for Affective Disorders (KSADS), and at 3-month follow up

SECONDARY OUTCOMES:
Change in Self-report Anxiety | Baseline and post-intervention (4 weeks), and at 3-month follow up.
  Change in self-report anxiety symptoms from baseline at 4-weeks on the Screen for Child Anxiety Related Disorders (SCARED), and at 3-month follow up.
Change in Dwell time on negative faces | Baseline and post-intervention (4 weeks), and at 3-month follow up.
  Change in dwell time on negative faces, from baseline at 4-weeks, using eye-tracking measures on a free-viewing attention task, and at 3-month follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No